CLINICAL TRIAL: NCT01273519
Title: Assessment of Pain Management in Rheumatoid Arthritis, Psoriatic Arthritis and Ankylosing Spondylitis Patients Who Are About to be Treated With Adalimumab
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Raffeiner GmbH (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P12-585
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Results first posted 2014-02-24 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-02

CONDITIONS: Rheumatoid Arthritis; Ankylosing Spondylitis; Psoriatic Arthritis
Keywords: Ankylosing; Rheumatoid; Antibodies; Arthritis; Pain; Antirheumatic Agents; Psoriatic; Spondylitis; Monoclonals
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylitis, Ankylosing; Arthritis, Psoriatic; Arthritis; Pain; Spondylitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- RA, PsA, AS: Participants with rheumatoid arthritis (RA), psoriatic arthritis (PsA) and ankylosing spondylitis (AS) prescribed Humira (adalimumab) in the usual manner and in accordance with the terms of the local marketing authorization with regards to dose, population and indication.

SUMMARY:
The purpose of this study is to assess whether or not adalimumab (Humira®) can influence pain medication in participants with rheumatoid arthritis (RA), psoriatic arthritis (PsA) and ankylosing spondylitis (AS) with or without comorbidities, which do not constitute a contraindication for adalimumab as stated in the released summary of product characteristics. Therefore it shall be evaluated if pain medication which is used in these participants is changed, reduced or stopped due to adalimumab treatment.

DETAILED DESCRIPTION:
This is a non-interventional, observational study in which Humira (adalimumab) is prescribed in the usual manner in accordance with the terms of the local marketing authorization with regards to dose, population and indication. The assignment of the patient to a Humira-containing regimen has to be decided in advance and has to be current practice. The prescription of Humira is clearly separated from the decision to include the participant in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years for rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis
* Patients must fulfill international and national guidelines for the use of a biological disease modifying antirheumatic drug in rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis (chest x-ray and interferon gamma release assay or purified protein derivative-skin test negative for tuberculosis). In addition one of the following criteria must be fulfilled:

  * unsatisfactory disease modifying antirheumatic drug response defined as failure to treatment with at least two disease modifying antirheumatic drugs including Methotrexate in patients with rheumatoid arthritis or psoriatic arthritis
  * unsatisfactory non steroidal antiinflammatory drug response in patients with ankylosing spondylitis or unsatisfactory response to prior biological disease modifying antirheumatic drugs in patients with rheumatoid arthritis or psoriatic arthritis or ankylosing spondylitis

Exclusion Criteria:

* Patients who meet contraindications as outlined in the latest version of the Humira syringe® summary of product characteristics and Humira Pen® summary of product characteristics
* Patients participating in another study program or clinical trial
* Patients who have been treated with Humira before

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary care clinic and medical practice specialized in rheumatology
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Dworan-Timler, MD, Study Director — AbbVie Austria
Locations (15):
- Austria (15):
  - Site Reference ID/Investigator# 52144, Bludenz
  - Site Reference ID/Investigator# 44915, Fürstenfeld
  - Site Reference ID/Investigator# 44910, Gloggnitz
  - Site Reference ID/Investigator# 44914, Graz
  - Site Reference ID/Investigator# 52143, Innsbruck
  - Site Reference ID/Investigator# 44916, Klagenfurt
  - Site Reference ID/Investigator# 44911, Linz
  - Site Reference ID/Investigator# 44912, Linz
  - Site Reference ID/Investigator# 44913, Linz
  - Site Reference ID/Investigator# 44906, Neudorf
  - Site Reference ID/Investigator# 44909, Sankt Pölten
  - Site Reference ID/Investigator# 52145, Spitz
  - Site Reference ID/Investigator# 44908, Stockerau
  - Site Reference ID/Investigator# 67062, Vienna
  - Site Reference ID/Investigator# 57304, Vöcklabruck

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Rheumatoid Arthiritis (RA): Participants with rheumatoid arthritis (RA) prescribed Humira (adalimumab) in the usual manner and in accordance with the terms of the local marketing authorization with regards to dose, population and indication.
- Psoriatic Arthritis (PsA): Participants with psoriatic arthritis (PsA) prescribed Humira (adalimumab) in the usual manner and in accordance with the terms of the local marketing authorization with regards to dose, population and indication.
- Ankylosing Spondylitis (AS): Participants with ankylosing spondylitis (AS) prescribed Humira (adalimumab) in the usual manner and in accordance with the terms of the local marketing authorization with regards to dose, population and indication.
Period: Overall Study
Arm/Group | Rheumatoid Arthiritis (RA) | Psoriatic Arthritis (PsA) | Ankylosing Spondylitis (AS)
Started | 78 | 30 | 47
Completed | 59 | 25 | 39
Not Completed | 19 | 5 | 8
Not completed — Adverse Event | 3 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 3
Not completed — Lack of Efficacy | 8 | 3 | 4
Not completed — Other | 6 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rheumatoid Arthiritis (RA) | Psoriatic Arthritis (PsA) | Ankylosing Spondylitis (AS) | Total
Number analyzed (Participants) | 78 | 30 | 47 | 155
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.76 (13.11) | 48.07 (12.71) | 42.02 (10.97) | 49.6 (13.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 9 | 18 | 94
  Male | 11 | 21 | 29 | 61

OUTCOME MEASURES:

1. Primary Outcome: Participant Assessment of Present Pain Intensity Recorded on a Visual Analogue Scale (VAS) at Baseline and Months 3, 6, 9, and 12
Description: Participants measured their present pain intensity on a visual analogue scale (VAS), where the responses were on a continuous range from 0 (no pain) to 100 (worst pain imaginable).
Time Frame: Baseline, Months 3, 6, 9, 12
Population: All participants with an assessment. n=number of participants with an assessment at time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RA, PsA, AS
Number analyzed (Participants) | 152
units on a scale
  Baseline, n=152 | 58.32 (22.01)
  Month 3, n=143 | 34.28 (24.74)
  Month 6, n=116 | 27.14 (22.69)
  Month 9, n=112 | 21.71 (20.21)
  Month 12, n=105 | 14.62 (16.88)

2. Primary Outcome: Physician Assessment of Present Pain Intensity Recorded on a Visual Analogue Scale (VAS) at Baseline and Months 3, 6, 9, and 12
Description: Physicians measured participants' present pain intensity on a visual analogue scale (VAS), where the responses were on a continuous range from 0 (no pain) to 100 (worst pain imaginable).
Time Frame: Baseline, Months 3, 6, 9, 12
Population: All participants with an assessment. n=number of participants with an assessment at time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RA, PsA, AS
Number analyzed (Participants) | 152
units on a scale
  Baseline, n=152 | 56.55 (21.57)
  Month 3, n=141 | 31.19 (23.95)
  Month 6, n=114 | 25.32 (22.13)
  Month 9, n=108 | 19.06 (18.46)
  Month 12, n=105 | 12.2 (15.1)

3. Primary Outcome: Participant Assessment of Present Pain Intensity Recorded on a Likert Scale at Baseline and Month 12
Description: Participants measured their present pain intensity by specifying their level of pain in response to the question "How intensive is your pain at present?" on a 4-point Likert scale, where 0 = no pain; 1 = mild pain, 2 = moderate pain, 3 = severe pain.
Time Frame: Baseline, Month 12
Population: All participants with an assessment at time point.
Measure: Number; unit: participants
Groups:
- RA, PsA, AS: Baseline: Participants at Baseline with rheumatoid arthritis (RA), psoriatic arthritis (PsA) and ankylosing spondylitis (AS) prescribed Humira (adalimumab) in the usual manner and in accordance with the terms of the local marketing authorization with regards to dose, population and indication.
- RA, PsA, AS: Month 12: Participants at Month 12 with rheumatoid arthritis (RA), psoriatic arthritis (PsA) and ankylosing spondylitis (AS) prescribed Humira (adalimumab) in the usual manner and in accordance with the terms of the local marketing authorization with regards to dose, population and indication.
Arm/Group | RA, PsA, AS: Baseline | RA, PsA, AS: Month 12
Number analyzed (Participants) | 150 | 105
participants
  No Pain | 4 | 49
  Mild Pain | 22 | 40
  Moderate Pain | 61 | 14
  Severe Pain | 63 | 2

4. Primary Outcome: Participant Assessment of Pain Intensity in the Past 3 Months Recorded on a Visual Analogue Scale (VAS) at Baseline and Months 3, 6, 9, and 12
Description: Participants measured their pain intensity in the past 3 months on a visual analogue scale (VAS), where the responses were on a continuous range from 0 (no pain) to 100 (worst pain imaginable).
Time Frame: Baseline, Months 3, 6, 9, 12
Population: All participants with an assessment. n=number of participants with an assessment at time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RA, PsA, AS
Number analyzed (Participants) | 150
units on a scale
  Baseline, n=150 | 64.31 (19.79)
  Month 3, n=142 | 38.24 (25.12)
  Month 6, n=114 | 30.89 (21.5)
  Month 9, n=109 | 24.74 (20.3)
  Month 12, n=105 | 17.36 (17.57)

5. Primary Outcome: Participant Assessment of Pain Intensity in the Past 3 Months Recorded on a Likert Scale at Baseline and Month 12
Description: Participants measured their pain intensity in the past 3 months by specifying their level of pain in response to the question "How intensive was your pain on average in the past 3 months?" on a 4-point Likert scale, where 0 = no pain; 1 = mild pain, 2 = moderate pain, 3 = severe pain.
Time Frame: Baseline, Month 12
Population: All participants with an assessment.
Measure: Number; unit: participants
Arm/Group | RA, PsA, AS: Baseline | RA, PsA, AS: Month 12
Number analyzed (Participants) | 150 | 105
participants
  No pain | 0 | 40
  Mild | 10 | 44
  Moderate | 71 | 19
  Severe | 69 | 2

6. Primary Outcome: Participant Assessment of the Pattern of Pain Progression (Daytime/Nocturnal) in the Past 3 Months at Baseline and Month 12
Description: Participants assessed the pattern of their pain progression in the past 3 months according to the following descriptors: intermittent (daytime and/or nocturnal); mostly daytime; mostly nocturnal; continuous (daytime and nocturnal).
Time Frame: Baseline, Month 12
Population: All participants with an assessment. n=number of participants with an assessment at time point.
Measure: Number; unit: participants
Arm/Group | RA, PsA, AS: Baseline | RA, PsA, AS: Month 12
Number analyzed (Participants) | 150 | 87
participants
  Intermittent | 41 | 42
  Mostly daytime | 18 | 22
  Mostly nocturnal | 26 | 13
  Continuous | 65 | 10

7. Primary Outcome: Participant Assessment of the Pattern of Pain Progression (Sudden/Creeping) in the Past 3 Months at Baseline and Month 12
Description: Participants assessed the pattern of their pain progression in the past 3 months according to the following descriptors: the type of beginning of pain was mostly sudden; the type of beginning of pain was mostly creeping.
Time Frame: Baseline, Month 12
Population: All participants with an assessment. n=number of participants with an assessment at time point.
Measure: Number; unit: participants
Arm/Group | RA, PsA, AS: Baseline | RA, PsA, AS: Month 12
Number analyzed (Participants) | 141 | 86
participants
  Sudden | 40 | 30
  Creeping | 101 | 56

8. Primary Outcome: Participant Assessment of the Presence of Nocturnal Pain Progression in the Past 3 Months at Baseline and Month 12
Description: Participants assessed how often on average they noted the presence of nocturnal pain in the past 3 month according to the following descriptors: never; rarely (not exceeding once a week), every night (awake from sleep at least once a night), more than once a night per week.
Time Frame: Baseline, Month 12
Population: All participants with an assessment.
Measure: Number; unit: participants
Arm/Group | RA, PsA, AS: Baseline | RA, PsA, AS: Month 12
Number analyzed (Participants) | 148 | 103
participants
  Never | 3 | 41
  Rarely | 14 | 42
  Every night | 57 | 3
  More than once a night per week | 74 | 17

9. Secondary Outcome: Mean Medical Outcomes Study Short Form 36 (SF-36) Summary of Scales at Baseline, and Months 3, 6, 9, and 12
Description: The SF-36 determines participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Items 1 to 4 primarily contribute to the physical component summary score (PCS) of the SF-36. Items 5 to 8 primarily contribute to the mental component summary score (MCS) of the SF-36. Scores on each item are summed and averaged (range = 0 [worst] to 100 [best ]). The standard recall period is 4 weeks. Increases from Baseline indicate improvement.
Time Frame: Baseline, Months 3, 6, 9, 12
Population: All participants with an assessment. n=number of participants with an assessment at time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RA, PsA, AS
Number analyzed (Participants) | 144
units on a scale
  Physical functioning: Baseline, n=143 | 46.9 (26.0)
  Physical functioning: Month 3, n=131 | 62.1 (28.9)
  Physical functioning: Month 6, n=104 | 66.9 (27.4)
  Physical functioning: Month 9, n=96 | 71.9 (25.9)
  Physical functioning: Month 12, n=94 | 77.1 (25.8)
  Role functioning physical: Baseline, n=142 | 16.7 (33.0)
  Role functioning physical: Month 3, n=129 | 42.4 (44.9)
  Role functioning physical: Month 6, n=103 | 48.8 (44.5)
  Role functioning physical: Month 9, n=96 | 54.7 (44.8)
  Role functioning physical: Month 12, n=93 | 63.4 (44.0)
  Bodily pain: Baseline, n=144 | 27.2 (19.0)
  Bodily pain: Month 3, n=131 | 52.1 (25.6)
  Bodily pain: Month 6, n=104 | 56.3 (24.1)
  Bodily pain: Month 9, n=96 | 62.8 (23.8)
  Bodily pain: Month 12, n=95 | 73.2 (23.2)
  General health: Baseline, n=141 | 38.3 (16.5)
  General health: Month 3, n=131 | 46.6 (19.8)
  General health: Month 6, n=104 | 49.9 (18.9)
  General health: Month 9, n=96 | 58.3 (20.8)
  General health: Month 12, n=95 | 64.9 (21.4)
  Vitality: Baseline, n=144 | 36.6 (18.9)
  Vitality: Month 3, n=131 | 51.3 (21.4)
  Vitality: Month 6, n=104 | 56.3 (21.6)
  Vitality: Month 9, n=96 | 61.4 (20.1)
  Vitality: Month 12, n=95 | 68.0 (18.7)
  Social functioning: Baseline, n=142 | 42.5 (23.8)
  Social functioning: Month 3, n=130 | 62.6 (25.4)
  Social functioning: Month 6, n=104 | 66.7 (25.1)
  Social functioning: Month 9, n=96 | 72.7 (23.7)
  Social functioning: Month 12, n=94 | 82.4 (19.9)
  Role functioning emotional: Baseline, n=143 | 38.0 (43.6)
  Role functioning emotional: Month 3, n=128 | 60.7 (45.7)
  Role functioning emotional: Month 6, n=103 | 61.2 (43.1)
  Role functioning emotional: Month 9, n=96 | 76.0 (39.8)
  Role functioning emotional: Month 12, n=95 | 85.6 (31.8)
  Mental health: Baseline, n=143 | 48.9 (18.5)
  Mental health: Month 3, n=131 | 63.0 (19.1)
  Mental health: Month 6, n=103 | 67.5 (19.7)
  Mental health: Month 9, n=94 | 72.1 (18.9)
  Mental health: Month 12, n=95 | 77.1 (18.0)

10. Secondary Outcome: Mean Health Assessment Questionnaire-Disability Index (HAQ-DI) Scores at Baseline, and Months 3, 6, 9, and 12
Description: The HAQ-DI is a participant-reported questionnaire. It consists of 20 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 to 3, where 0 represents no disability and 3 represents very severe, high-dependency disability. The minimal clinically important difference defined for the HAQ-DI is ≥0.22. HAQ remission, indicating normal physical function, is defined as HAQ-DI < 0.5.
Time Frame: Baseline, Months 3, 6, 9, 12
Population: All participants with an assessment. n=number of participants with an assessment at time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rheumatoid Arthiritis (RA) | Psoriatic Arthritis (PsA) | Ankylosing Spondylitis (AS)
Number analyzed (Participants) | 73 | 28 | 6
units on a scale
  Baseline, n=73, 28, 6 | 1.31 (0.69) | 0.85 (0.57) | 0.88 (0.62)
  Month 3, n=66, 26, 2 | 0.94 (0.72) | 0.62 (0.64) | 0.75 (0.35)
  Month 6, n=53, 19, 0 | 0.87 (0.78) | 0.77 (0.69) | NA (NA) — no participants had an assessment at this time point
  Month 9, n=46, 21, 0 | 0.83 (0.71) | 0.54 (0.54) | NA (NA) — no participants had an assessment at this time point
  Month 12, n=48, 22, 0 | 0.68 (0.72) | 0.51 (0.57) | NA (NA) — no participants had an assessment at this time point

11. Secondary Outcome: Mean Rheumatoid Arthritis Disease Activity Index (RADAI) at Baseline, and Months 3, 6, 9, and 12
Description: The RADAI is a questionnaire for patients used for measuring disease activity. The index consists of 6 questions. The items ask the participants about (1) global disease activity in the last 6 months, (2) disease activity in terms of current swollen and tender joints, (3) arthritis pain, (4) the current status of health, (5) duration of morning stiffness and (6) tender joints to be rated in a joint list. The joint list asks about pain in the left and right shoulders, elbows, wrists, fingers, hips, knees, ankles and toes. The first 4 items are all rated on a numeric rating scale from 0 to 10, where higher scores indicate more disease activity. The scores on the last 2 items range from 0 to 6 and 0 to 48, respectively, but are transformed on the same scale of 0 to 10. The RADAI total score is the sum of individual items divided by 5 (range 0-10), with a higher score signifying more disease activity.
Time Frame: Baseline, Months 3, 6, 9, 12
Population: All participants with an assessment. n=number of participants with an assessment at time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rheumatoid Arthiritis (RA) | Psoriatic Arthritis (PsA) | Ankylosing Spondylitis (AS)
Number analyzed (Participants) | 72 | 27 | 5
units on a scale
  Baseline, n=72, 27, 5 | 5.46 (1.6) | 4.72 (1.69) | 4.61 (2.57)
  Month 3, n=67, 22, 2 | 3.78 (2.14) | 2.41 (1.63) | 4.23 (2.15)
  Month 6, n=53, 18, 0 | 2.74 (2.1) | 2.34 (2.06) | NA (NA) — no participants had an assessment at this time point
  Month 9, n=46, 20, 0 | 2.19 (1.81) | 1.81 (1.86) | NA (NA) — no participants had an assessment at this time point
  Month 12, n=49, 21, 0 | 1.72 (1.83) | 1.55 (1.91) | NA (NA) — no participants had an assessment at this time point

12. Secondary Outcome: Mean Bath Ankylosing Spondylitis Functional Index (BASFI) Scores at Baseline, and Months 3, 6, 9, and 12
Description: The BASFI is a set of 10 questions designed to determine the degree of functional limitation in those with AS. The 10 questions were chosen with a major input from patients with AS. The first 8 questions consider activities related to functional anatomy. The final 2 questions assess the participants' ability to cope with everyday life. A visual analogue scale (with 0 being "easy" and 10 "impossible") is used to answer the questions on the test.
Time Frame: Baseline, Months 3, 6, 9, 12
Population: Participants with AS or PsA and an assessment. n=number of participants with an assessment at time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- PsA, AS: Participants with psoriatic arthritis (PsA) and ankylosing spondylitis (AS) prescribed Humira (adalimumab) in the usual manner and in accordance with the terms of the local marketing authorization with regards to dose, population and indication.
Arm/Group | PsA, AS
Number analyzed (Participants) | 72
units on a scale
  Baseline, n=72 | 5.46 (1.6)
  Month 3, n=67 | 3.78 (2.14)
  Month 6, n=53 | 2.74 (2.1)
  Month 9, n=46 | 2.19 (1.81)
  Month 12, n=49 | 1.72 (1.83)

13. Secondary Outcome: Mean Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) for Participants With Ankylosing Spondylitis (AS) at Baseline, and Months 3, 6, 9, and 12
Description: The BASDAI is used for measuring and evaluating disease activity in AS. This index consists of 6 questions pertaining to the 5 major symptoms of AS: fatigue, spinal pain, joint pain/swelling, areas of localized tenderness (or enthesitis, defined as inflammation of tendons and ligaments), duration of morning stiffness, severity of morning stiffness. A visual analogue scale ranging from 0 (none) to 10 (very severe) is used to answer the questions. The final BASDAI score averages the individual assessments for a final score range of 0-10 (0 being no problem and 10 being the worst problem).
Time Frame: Baseline, Months 3, 6, 9, 12
Population: All participants with an assessment. n=number of participants with an assessment at time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ankylosing Spondylitis (AS)
Number analyzed (Participants) | 45
units on a scale
  Baseline, n=45 | 5.65 (2.25)
  Month 3, n=44 | 3.24 (2.25)
  Month 6, n=39 | 2.62 (2.55)
  Month 9, n=34 | 1.97 (2.15)
  Month 12, n=32 | 1.23 (1.9)

14. Secondary Outcome: Mean Erythrocyte Sedimentation Rate (ESR) at Baseline, and Months 3, 6, 9, and 12
Description: The ESR is a practicable and sensitive but not specific parameter for measuring disease progression. By means of the ESR it can be generally distinguished between an active and nonactive rheumatic disease. The normal reference range is, as a rule, 0 to 10 mm/h for men and 0 to 15 mm/h for women. The higher the ESR value out of the normal range, the higher is the disease activity.
Time Frame: Baseline, Months 3, 6, 9, 12
Population: All participants with an assessment. n=number of participants with an assessment at time point.
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | Rheumatoid Arthiritis (RA) | Psoriatic Arthritis (PsA) | Ankylosing Spondylitis (AS)
Number analyzed (Participants) | 69 | 25 | 40
mm/h
  Baseline, n=69, 25, 40 | 32.87 (17.89) | 23.96 (19.41) | 28.58 (22.87)
  Month 3, n=68, 25, 40 | 21.95 (18.25) | 13.4 (15.05) | 12.45 (10.33)
  Month 6, n=58, 21, 37 | 21.98 (19.22) | 14.81 (16.62) | 13.24 (10.29)
  Month 9, n=51, 23, 33 | 25.49 (22.45) | 14.09 (16.9) | 12.79 (7.75)
  Month 12, n=49, 21, 30 | 19.94 (19.63) | 13.33 (15.32) | 12.0 (7.95)

15. Secondary Outcome: Mean C-reactive Protein (CRP) at Baseline, and Months 3, 6, 9, and 12
Description: The CRP is an acute phase reactant plasma protein, normally produced by the liver, which is commonly used as an indirect measure of the extent and activity of an inflammation. The CRP normal reference range in the blood is, as a rule, from 0 to 1.0 mg/dL.
Time Frame: Baseline, Months 3, 6, 9, 12
Population: All participants with an assessment. n=number of participants with an assessment at time point.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Rheumatoid Arthiritis (RA) | Psoriatic Arthritis (PsA) | Ankylosing Spondylitis (AS)
Number analyzed (Participants) | 57 | 21 | 39
mg/dL
  Baseline, n=57, 21, 39 | 1.83 (2.65) | 1.56 (3.25) | 1.18 (1.69)
  Month 3, n=61, 22, 39 | 4.3 (10.88) | 2.31 (7.39) | 0.84 (1.89)
  Month 6, n=50, 17, 35 | 1.95 (4.03) | 1.25 (1.94) | 1.57 (3.14)
  Month 9, n=44, 17, 32 | 2.16 (3.85) | 5.33 (12.96) | 1.14 (2.35)
  Month 12, n=45, 18, 31 | 1.73 (3.89) | 2.42 (5.36) | 1.26 (3.31)

16. Primary Outcome: Participant Assessment of the Presence of Distress Caused by Pain in the Last 3 Months Recorded on a Likert Scale at Baseline and Month 12
Description: Participants indicated their perception of average distress caused by pain in the past 3 months on a 5-point Likert scale, where; 0 = no pain, 1 = not distressed, 2 = slightly distressed, 3 = moderately distressed, 4 = greatly distressed by pains.
Time Frame: Baseline, Month 12
Population: All participants with an assessment.
Measure: Number; unit: participants
Arm/Group | RA, PsA, AS: Baseline | RA, PsA, AS: Month 12
Number analyzed (Participants) | 150 | 104
participants
  No pain | 0 | 33
  Not distressed by pain | 0 | 23
  Slightly distressed by pain | 10 | 28
  Moderately distressed by pain | 71 | 18
  Greatly distressed by pain | 69 | 2

ADVERSE EVENTS:
Time Frame: All serious adverse events were reported from the time of informed consent (and adverse events were reported from Baseline) until 70 days following the intake of the last dose of physician-prescribed treatment. Duration of study was 871 days.
Arm/Group | RA, PsA, AS
Serious Adverse Events (participants affected / at risk) | 3/155
Other Adverse Events (participants affected / at risk) | 21/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RA, PsA, AS (N=155)
Carotid artery stenosis (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Respiratory tract infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Treatment failure (General disorders) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RA, PsA, AS (N=155)
Drug ineffective (Immune system disorders) | 17
Sleep disorder (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1
Intervetebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Arthritis reactive (Infections and infestations) | 1
C-reactive protein increased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.